CLINICAL TRIAL: NCT05374655
Title: A Multicenter Randomized Controlled Clinical Study of Preoperative Glycosylated Hemoglobin Control Strategies on the Effectiveness of Cox-Maze IV Procedure for Atrial Fibrillation During Cardiac Surgery
Brief Title: Outcomes Study of Glycosylated Hemoglobin Control in Cox-Maze IV During Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kun Hua (Other)
Collaborators: Peking University People's Hospital (Other); Peking University International Hospital (Other); Beijing Huaxin Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Kun Hua, Deputy Chief Surgeon, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: blank
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Cardiac Surgery
Keywords: Cardiac Surgery; Atrial Fibrillation; Glycosylated Hemoglobin; Cox-Maze IV
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative blood glucose control (Experimental): Under the guidance of endocrinologists, the patient's hypoglycemic strategy is formulated, follow-up guidance is guided by the patient to take the drug, the HbA1c level is reviewed after 6 weeks, the preoperative HbA1c < 7.5% is performed surgically, and if it is still above the standard, the hypoglycemic therapy is continued, during which the patient is administered according to the corresponding heart disease type.
  Interventions: Other: Preoperative blood glucose control
- Preoperative blood glucose uncontrol (No Intervention): Patients included in this group ≥ 7.5% preoperative HbA1c and underwent surgery directly

INTERVENTIONS:
Other: Preoperative blood glucose control — Patients included in this group, under the guidance of endocrinologists, develop hypoglycemic strategies for patients, follow up and guide patients to take medication, review HbA1c levels after 6 weeks, perform surgical treatment if they meet preoperative HbA1c<7.5%, continue hypoglycemic therapy if still above standards, and administer drugs according to the corresponding type of heart disease during this period.
  Arms: Preoperative blood glucose control

SUMMARY:
In recent years, a growing body of research has shown that diabetes plays an important role in the development and recurrence of atrial fibrillation. How to achieve the treatment and prevention of recurrence of atrial fibrillation through appropriate blood glucose control is the current focus of clinical research. Glycosylated hemoglobin (HbA1c) is the product of a non-enzymatic reaction in which hemoglobin in red blood cells is combined with sugars in the serum (mainly glucose). The purpose of this multicenter, randomized controlled study is to compare the effects of different glycosylated hemoglobin control strategies on the effectiveness of Cox-Maze IV procedure for atrial fibrillation during cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Elective cardiac surgery
* A clear diagnosis of diabetes mellitus, and HbA1c ≥ 7.5% at the time of initial diagnosis and treatment
* Preoperative combination of persistent or long-term persistent atrial fibrillation

Exclusion Criteria:

* Emergency surgery or limited-term surgery
* Previous cardiac surgery
* Left atrial diameter > 65 mm
* Serum creatine > 1.8 mg/dL
* Previous severe liver disease
* Pregnant or planning to become pregnant
* Have a malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of atrial fibrillation recurrence | one year post operative
  Atrial fibrillation heart rate recorded on a 24-hour Holter electrocardiogram persisted for more than 30 seconds

SECONDARY OUTCOMES:
Rate of atrial fibrillation recurrence | 6 months post operative
  Atrial fibrillation heart rate recorded on a 24-hour Holter electrocardiogram persisted for more than 30 seconds
All-cause Mortality | one year post operative
  All-cause mortality identified during one-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kun Hua, Study Chair — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China